CLINICAL TRIAL: NCT02951377
Title: Mechanical Diagnosis and Treatment and/or Transforaminal Epidural Steroid Injections Versus Usual Care for Chronic Lumbar Radiculopathy: A Pilot Study.
Brief Title: Mechanical Diagnosis and Treatment and/or Steroid Injections for Lumbar Radiculopathy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruitment
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other); Alberta College and Association of Phyiotherapists (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RES0032934
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2020-03

CONDITIONS: Sciatica; Lumbosacral Radiculopathy; Lumbar Disc Rupture
Keywords: mechanical diagnosis therapy (MDT); physical therapy; steroid injection; exercise
MeSH Terms: conditions — Sciatica; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Wait list control - usual care - free to pursue other treatments prescribed by the patients family physician
- MDT +/- TESI (Experimental): Exercise (MDT approach) and/or Transforaminal epidural steroid injection (20mg dexamethasone 0.5cc lidocaine 2%). Patients will further classified into centraliser (group 2a) and non-centralising pain responses (group 2b). Group 2a: will continue with exercise (MDT approach). Group 2b: Patients with a non-centralising pain response will be offered Transforaminal epidural steroid injection (20mg dexamethasone 0.5cc lidocaine 2%), under fluoroscopic guidance with contrast medium (Omni Pac 240). Two weeks after completion of the MDT or TESI intervention, patients will be reassessed and treated consistent with their response: 1) resolved: advice on remaining active; 2) centralising: daily exercises based on MDT principles; 3) non-centralising but significant less pain: advice to remain active, with respect for worsening leg pain; and 4) persisting high levels of pain and/or disability: advise to remain active as tolerated and consult family physician.
  Interventions: Other: Exercise (MDT approach); Drug: Transforaminal epidural steroid injection (20mg dexamethasone 0.5cc lidocaine 2%)

INTERVENTIONS:
Other: Exercise (MDT approach) — Postural or movement exercises of the lower back that aim to centralise and reduce pain intensity.
  Arms: MDT +/- TESI
Drug: Transforaminal epidural steroid injection (20mg dexamethasone 0.5cc lidocaine 2%) — An epidural steroid injection (20mg dexamethasone 0.5cc lidocaine 2%), under guidance of fluoroscopy is used to reduce inflammation at a lumbar spinal nerve root(s).
  Arms: MDT +/- TESI

SUMMARY:
Aim 1: The primary aim of this study is to test the feasibility of Mechanical Diagnosis and Treatment (MDT) +/- transforaminal epidural steroid injections (TESI) on pain and disability in patients awaiting physiatry consult for lumbar radiculopathy secondary to lumbar disc herniation, compared to usual care within the current healthcare system in Calgary, Alberta, Canada.

Hypothesis: the investigators hypothesise that centralisers treated with MDT and non-centralisers receiving TESIs + MDT will have demonstrate reductions in self-reported pain and disability, compared to usual care controls.

Aim 2: the investigators will also describe the potential impact on healthcare resources by tracking surgical rates and self-reported healthcare utilisation during the study period.

Hypothesis: based on predicted reductions in pain and disability, the investigators hypothesise that there will be a trend toward overall less healthcare utilisation (including surgery) in the MDT guided group compared to the surgical wait list group.

DETAILED DESCRIPTION:
Study Purpose and Specific Objectives: This pilot study aims to determine the feasibility of conducting a definitive clinical trial of MDT +/- TESI in patients awaiting physiatry consult for lumbar radiculopathy secondary to lumbar disc herniation compared to usual care.

Research Design and Methodology:

Design and participants: Randomised clinical trial pilot study. Eligible candidates will be identified by Physiatrists at a Physiatry clinic in Calgary. The investigators will recruit 30 patients (15 per group). Fifteen - twenty subjects per group provide reasonable bias-corrected estimates for medium effects. Inclusion criteria: Leg dominant pain secondary to lumbar disc protrusion confirmed on MRI with duration > 3 months, at least one neurological sign and able to speak English and provide written informed consent. Exclusion criteria: pregnancy and specific causes of low back pain (LBP) not directly related to herniated discs, progressive neurological signs and/or cauda equine syndrome, or contraindication for the use of corticosteroids or fluoroscopy. Consecutive patients will randomised into either the intervention described below to enable an estimation of the magnitude of the treatment effect or the usual care will be followed to estimate the magnitude of effect for the control group.

Interventions: Group 1- Control group: Outcome assessments will be conducted on patients on the wait list for physiatry consultation at baseline, 6 weeks, and 3 months. Group 2 - Intervention group (MDT group): Consistent with the MDT approach, patients will be initially assessed for centralisation over 2 visits by a Credentialed MDT therapist and further classified into centraliser (group 2a) and non-centralising pain responses (group 2b). A centralising pain response is defined as those whose most distal pain is reduced and retreats toward mid-line (e.g., pain now above knee) in response to certain postures and repeated end-range movement testing. Group 2a, Centralisers: Patients with a centralising pain response will continue with treatment based on MDT principles and will complete an exercise diary to indicate the frequency in which the exercises were performed daily. Group 2b, Non-centralisers: Patients with a non-centralising pain response will be offered TESIs followed by MDT. TESIs of 20mg dexamethasone and 0.5cc lidocaine 2%, under fluoroscopic guidance with contrast medium (Omni Pac 240) as described by the Spine Intervention Society (SIS) guidelines will be provided. Segment level will be determined based on MRI findings in combination with the clinical examination findings.

Two weeks after completion of the MDT or TESI intervention, patients will be reassessed and treated in a manner consistent with their presenting pain response classification: 1) resolved: advice on remaining active; 2) centralising: treated according to MDT principles with direction specific exercises and postural advise; 3) non-centralising but significant less pain: advice to remain active, with respect for worsening leg pain; and 4) persisting high levels of pain and/or disability: advise to remain active as tolerated and consult family physicians. Those who continue to perform MDT exercises will complete an exercise diary to indicate the frequency in which the exercises were performed daily

Outcome assessments: Assessing and treating therapists are credentialed in MDT and will be blinded to outcomes. The following outcomes will be assessed in all groups at baseline, 6 weeks, and 3 months. The primary outcome measures will be the Roland-Morris Disability Questionnaire (RMDQ) adapted and validated for sciatica, leg pain intensity, and global perceived effect (GPE). Average leg pain intensity will be measured using a numeric rating scale ranging from 0 (no pain) to 10 (worst imaginable pain) over the past 24 hours. GPE will be measured using a 7 point Likert scale, with lower scores suggesting recovery and higher scores suggesting worsening. Secondary outcome measures will include fear avoidance (FABQ), general health (SF-12), and medication use. Demographics will also be collected. In addition, participants who are prescribed exercises will complete a diary indicating the frequency at which the exercises were performed.

Data analysis: Leg pain intensity at 3 months, measured using a 10 point numeric rating scale (NRS) will be the primary outcome for which the larger more definitive study will be planned. An independent t-test will be used to estimate the effect sizes of the intervention group compared to the control group. Independent t-tests will also be applied to the other outcome measures for exploratory purposes. Statistical significance will be set at α=0.05. Descriptive statistics will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* leg dominant pain secondary to lumbar disc protrusion confirmed on MRI with duration > 3 months, at least one neurological sign and able to speak English and provide written informed consent.

Exclusion Criteria:

* Pregnancy and specific causes of LBP not directly related to herniated discs, progressive neurological signs and/or cauda equine syndrome, or contraindication for the use of corticosteroids or fluoroscopy. These features primarily represent patients who are not suitable for the interventions offered in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Roland-Morris Disability Questionnaire | 3 months after baseline
Leg pain intensity numeric rating scale | 3 months after baseline
Global rating of change in the condition | 3 months after baseline
  Global perceived effect: measured using a 7-point Likert scale asking patients how much their condition has improved/deteriorated since the start of the study.

SECONDARY OUTCOMES:
Fear avoidance beliefs questionnaire | 3 months after baseline
SF-12 general health | 3 months after baseline
Medication use | 3 months after baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Buenavista Physiotherapy, Calgary, Alberta, Canada